CLINICAL TRIAL: NCT06112470
Title: Alleged Drug Allergies in Military General Medicine: Patients' Experiences and Beliefs (ALLMED)
Brief Title: Alleged Drug Allergies in Military General Medicine: Patients' Experiences and Beliefs
Acronym: ALLMED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PPRC02
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Allergy Penicillin
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interview: Monocentric qualitative study with a descriptive socio-demographic section, a descriptive qualitative section on the experience and perception of allergy, then on the obstacles to allergological assessment, and finally a descriptive quantitative section to evaluate knowledge of antibiotic therapy.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Semi-structured interview on experiences, perceptions, beliefs and knowledge of drug allergy and barriers to allergological testing, with a view to content analysis.

SUMMARY:
This study focuses on the experience of the military patient reporting a suspected drug allergy, with its own specificities. Suspicions of drug allergies during a mission expose the doctor to difficulties.

This study will improve understanding of the allergy patient's point of view. The end result could be a set of ideas for measures to raise awareness among these patients, and motivate them to undergo an allergological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Military personnel (active or reservist)
* Reporting a drug allergy during a periodic medical check-up or during a consultation in a medical unit
* Not opposed to participating in the study.

Exclusion Criteria:

* Candidate on admission visit
* Opposition to study
* Minor (under 18 years of age)
* Pregnant, parturient or breast-feeding woman
* Person deprived of liberty by a judicial or administrative decision, person under psychiatric care
* Non-French nationals
* Person of full age subject to a legal protection measure
* Person unable to express non-opposition

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Military personnel reporting a drug allergy to antibiotics
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Patients' experiences of drug allergies | Through study completion (12 months)
  describe patients' experiences, perceptions, beliefs and knowledge of drug allergies in general practice in the army

SECONDARY OUTCOMES:
Patients' obstacles | Through study completion (12 months)
  describe the obstacles to allergological assessment

CONTACTS AND LOCATIONS:
Locations (1):
- 15ème antenne médicale - Camp des Matelots, Versailles, France

IPD SHARING:
Plan to Share IPD: Undecided